CLINICAL TRIAL: NCT04660487
Title: Relationship Between the Utilization and Degradation Rate of "FODMAPs" by Intestinal Flora and "GVHD"
Brief Title: Relationship Between "FODMAPs" and "GVHD"
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Qi Xiao-Fei, Dean, The First Affiliated Hospital of Soochow University
Other Study IDs: FODMAPS202001
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — intestinal flora
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the stem cell transplanting increasing, patients which effected with "GVHD" were also increased. To evaluation the relationship between "FODMAPs" and "GVHD", Bone marrow transplant patients were recruited.

DETAILED DESCRIPTION:
The feces were collected from the patients who had been successfully transplanted after bone marrow transplantation. After 24 hours of culture in the culture medium, the degradation rate of "FODMAPs" was detected, and the relationship between the degradation rate and the occurrence time and degree of "GVHD" was observed

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of "AML","ALL","MDS" or "MM" Disease;
2. Must be treated with bone marrow transplantation;
3. The transplanted bone marrow was successfully planted

Exclusion Criteria:

1. Gastrointestinal diseases；
2. Age>60; or Age<10；
3. Probiotics or prebiotics were taken before enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Successful bone marrow colonization after bone marrow transplantation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of GVHD | 90 days
  The occurrence time and degree of GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, Study Chair — SOOCHOW UNIV
Locations (1):
- 中国, Suzhou, Jiangsu, China